CLINICAL TRIAL: NCT01188486
Title: Pulmonary Interstitial Lymphography in Early Stage Lung Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Business decision
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Billy W. Loo Jr., Associate Professor of Radiation Oncology, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: IRB-18395; LUN0040 (Other: OnCore)
Record Dates: First submitted 2010-08-23; First posted 2010-08-25 (Estimated); Last update posted 2018-04-17 (Actual); Status verified 2018-04

CONDITIONS: Lung Cancer; Lung Cancer Non-Small Cell Cancer (NSCLC); Lung Cancer Small Cell Lung Cancer (SCLC); Mesothelioma
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma; Mesothelioma | interventions — Radiosurgery; Iohexol; iodixanol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- pulmonary interstitial lymphography (Experimental): stereotactic body radiation therapy & pulmonary interstitial lymphography
  Interventions: Radiation: Stereotactic Body Radiation Therapy (SBRT); Radiation: Computed Tomography (CT); Device: Cyberknife; Device: Trilogy; Device: True Beam; Drug: Iohexol; Drug: Iodixanol

INTERVENTIONS:
Radiation: Stereotactic Body Radiation Therapy (SBRT) — Standard of care diagnostic radiotherapy procedure
Radiation: Computed Tomography (CT) — For each participant, 3 chest CT scans will be obtained, 1 before and 2 after interstitial injection of the water-soluble contrast
Device: Cyberknife — Linear accelerator for producing high energy x-rays for radiation therapy.
Device: Trilogy — Linear accelerator for producing high energy x-rays for radiation therapy.
Device: True Beam — Linear accelerator for producing high energy x-rays for radiation therapy.
Drug: Iohexol — Aqueous solution of a nonionic, water-soluble radiographic contrast medium in prefilled cartridges with a molecular weight of 821.14 (iodine content 46.36%), available at 140, 180, 240, 300, and 350 mgI/mL.
  Other Names: Omnipaque; Omnipaque in Rediflo prefilled cartridges; Bis(2,3-dihydroxypropyl)-5-[N-(2,3-dihydroxypropyl)-acetamido]-2,4,6-triiodoisophthalamide
Drug: Iodixanol — Aqueous solution of a nonionic, water-soluble, dimeric, isosmolar, radiographic contrast medium with a molecular weight of 1550.20 (iodine content 49.1%), available in 2 concentrations, (270 mgI/mL and 320 mgI/mL.
  Other Names: Visipaque; 5,5´-[(2-hydroxy-1,3-propanediyl)bis (acetylimino)] bis[N,N´-bis(2,3-dihydroxypropyl)-2,4,6- triiodo-1,3- benzenedicarboxamide]

SUMMARY:
The stereotactic body radiation therapy (SBRT) procedure is an emerging alternative to the standard treatment for early stage non-small cell lung cancer (NSCLC), typically lobectomy with lymphadenectomy. This procedure (lobectomy) does not fulfill the medical need as many patients are poor operative candidates or decline surgery.

This study assesses the feasibility of stereotactic body radiation therapy (SBRT) as a tool to produce therapeutically useful computed tomography (CT) scans, using standard water-soluble iodinated compounds as the contrast agents.

DETAILED DESCRIPTION:
Non-small cell lung cancer (NSCLC) is the most deadly cancer in the world. NSCLC annually causes 150,000 deaths in the US and greater than 1 million worldwide. The standard treatment for early stage NSCLC is lobectomy with lymphadenectomy. However, many patients are poor operative candidates or decline surgery. An emerging alternative is Stereotactic Body Radiation Therapy (SBRT). Mounting evidence from phase 1-2 studies demonstrates that SBRT offers excellent local control. Most SBRT trials focused on small, peripheral tumors in inoperable patients. Increasingly, clinical trials study SBRT in operable patients, often with larger, central tumors.

Using clinical staging, a significant proportion of patients harbor occult nodal metastases when undergoing SBRT to the primary tumor alone. Subgroups of patients carry even higher risk of nodal metastases. These nodal metastases frequently would be removed by surgical intervention. However, SBRT, at present, is only directed at the primary tumor, potentially leading to regional failures in otherwise curable patients. To increase the effectiveness of SBRT for lung tumors, the next logical step is to explore whether the highest risk areas of disease spread can be identified and targeted. Regional failure could be reduced and outcome improved in a significant proportion of patients treated with SBRT if the primary nodal drainage (PND) were identified, targeted and treated in addition to the primary tumor.

We propose to conduct a study to determine the feasibility of visualizing, by computed tomography (CT) scans, water-soluble iodinated contrast materials after direct injection into the tumor. Integration into radiation therapy treatment planning may also be assessed.

ELIGIBILITY:
INCLUSION CRITERIA

* Either:

  * Established primary lung cancer/ cancer metastatic to lung, OR
  * Lesion suspicious for malignancy in lung, according to the following criteria:

    * Histopathologically confirmed lung cancer or cancer metastatic to lung, OR
    * Plan for biopsy of suspicious lung mass based on imaging (growth on serial CT scan or nodule/mass with focal hypermetabolism on FDG-PET scan), OR
    * Known metastatic cancer, with metastases to the lung based on imaging
* Age > 18 years old
* Eastern Clinical Oncology Group (ECOG) performance status 0, 1 or 2 (Appendix IV)
* No prior surgery, chemotherapy, or radiation for the current lung tumor

EXCLUSION CRITERIA

* Prior radiotherapy to thorax
* Iodine allergy
* Contraindication to receiving radiotherapy, unless undergoing surgery
* Pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2010-08; Primary Completion 2017-04-30 (Actual); Study Completion 2017-04-30 (Actual)

PRIMARY OUTCOMES:
- Feasibility and safety of identification of primary nodal drainage for purpose of radiation therapy targeting | 15 months

SECONDARY OUTCOMES:
- Feasibility of incorporating primary nodal drainage into radiation therapy planning process | 15 months

CONTACTS AND LOCATIONS:
Overall Officials: Billy W Loo, Jr, MD, PhD, Principal Investigator — Stanford University; Jonathan Abelson, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No